CLINICAL TRIAL: NCT02876783
Title: Analysis of Stroke Rehabilitation Outcomes
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1112012072
Record Dates: First submitted 2016-08-11; First posted 2016-08-24 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observational - No intervention

SUMMARY:
Observe and describe the relationships between impairments and function, systematically characterize recovery patterns and examine short and long term rehabilitation outcomes. This project is purely observational, descriptive and non-experimental. N=273

DETAILED DESCRIPTION:
This project involves an interdisciplinary stroke database of demographic variables and clinical measures collected during routine acute care, inpatient rehabilitation admission and discharge as well as follow up questionnaires at 6 month and 12 months to examine stroke recovery.

Our aim is to observe and describe the relationships between impairments and function, systematically characterize recovery patterns and examine short and long term rehabilitation outcomes.

This project is purely observational, descriptive and non experimental. No rehabilitation interventions or treatment procedures are being introduced, modified or studied.

ELIGIBILITY:
Inclusion Criteria:

Patients who have a confirmed primary diagnosis of cerebrovascular accident (CVA) as per radiological assessment, met the criteria to be admitted onto Baker 17 (the New York Presbyterian inpatient rehabilitation unit), and were administered standardized assessments or rating scales as part of routine standard care will be included in the database.

Exclusion Criteria:

Persons with stroke who could not be given standard assessments or rating scales (eg.

due to fatigue, decreased attention span, global aphasia or refusal) will not be included in data analysis.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only inpatients with a primary diagnosis of stroke who have been admitted to the inpatient rehabilitation unit (IRU) will be recruited for this study. Participants are medically stable (criteria for admission to the IRU) and have recently had a stroke.
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2012-07-25 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2017-01-03 (Actual)

PRIMARY OUTCOMES:
Participation questionnaire - Boston University Activity Measure for Post-Acute Care (AM-PAC) - administered by research assistant | 6 months
  Boston University Activity Measure for Post-Acute Care (AM-PAC) - A questionnaire that examines a set of functional activities that are likely to be encountered by most adults during daily routines within the context of either an inpatient episode of care or outpatient post acute services. AM-PAC item banks are organized into three functional areas: Basic Mobility (101 items), Daily Activity (70 items), and Applied Cognitive (69 items).
Participation questionnaire - Community Participation Indicators (CPI) - administered by research assistant | 6 months
  Community Participation Indicators (CPI) - Part 1 has the patient rate the frequency at which he/she does various activities, and asks if the activity is important to the patient. Part 2 has the patient rate how frequently their behavior aligns with various prompts, for example "I live my life the way that I want".
Participation questionnaire - Stroke Impact Scale (SIS) Participation domain - administered by research assistant | 6 months
  Stroke Impact Scale (SIS) Participation domain - A stroke-specific, self-reported, health status measure separated into 8 domains. We only administer the Participation domain.
Participation questionnaire - Boston University Activity Measure for Post-Acute Care (AM-PAC) - administered by research assistant | 12 months
  Boston University Activity Measure for Post-Acute Care (AM-PAC) - A questionnaire that examines a set of functional activities that are likely to be encountered by most adults during daily routines within the context of either an inpatient episode of care or outpatient post acute services. AM-PAC item banks are organized into three functional areas: Basic Mobility (101 items), Daily Activity (70 items), and Applied Cognitive (69 items).
Participation questionnaire - Community Participation Indicators (CPI) - administered by research assistant | 12 months
  Community Participation Indicators (CPI) - Part 1 has the patient rate the frequency at which he/she does various activities, and asks if the activity is important to the patient. Part 2 has the patient rate how frequently their behavior aligns with various prompts, for example "I live my life the way that I want".
Participation questionnaire - Stroke Impact Scale (SIS) Participation domain - administered by research assistant | 12 months
  Stroke Impact Scale (SIS) Participation domain - A stroke-specific, self-reported, health status measure separated into 8 domains. We only administer the Participation domain.
Mobility - Trunk Control Test - administered by physical therapist | Discharge (within 72 hours prior to discharge from inpatient rehabilitation unit - IRU)
  Includes four items: rolling to weak side, rolling to strong side, sitting up from lying down, balance in sitting position. Total score range 0-100
Mobility - Berg Balance Scale - administered by physical therapist | Discharge (within 72 hours prior to discharge from inpatient rehabilitation unit - IRU)
  Measures balance in patients by assessing performance of functional tasks. Total score range 0 (lowest level) to 56 (highest level)
Mobility - Timed Up and Go (TUG) - administered by physical therapist | Discharge (within 72 hours prior to discharge from inpatient rehabilitation unit - IRU)
  Assesses mobility, balance, walking ability and fall risk. Measured in seconds.
Mobility - Functional Reach Test - administered by physical therapist | Discharge (within 72 hours prior to discharge from inpatient rehabilitation unit - IRU)
  Measures maximum distance an individual can reach forward while standing in a fixed position.
Mobility - Postural Assessment Scale for Stroke (PASS) - administered by physical therapist | Discharge (within 72 hours prior to discharge from inpatient rehabilitation unit - IRU)
  A 12 item scale used for assessing postural control following stroke.
Mobility - 2 or 6 Minute Walk Test - administered by physical therapist | Discharge (within 72 hours prior to discharge from inpatient rehabilitation unit - IRU)
  Assesses patient's walking distance
Mobility - 10 Meter Walk Test - administered by physical therapist | Discharge (within 72 hours prior to discharge from inpatient rehabilitation unit - IRU)
  Assesses patient's walking speed
Mobility - Lower Extremity Motricity Index - administered by physical therapist | Discharge (within 72 hours prior to discharge from inpatient rehabilitation unit - IRU)
  Lower Extremity Motricity Index - Measures muscle strength of paretic side, post-stroke. Includes three items: ankle dorsiflexion, knee extension, hip flexion. Total score range 0-100
Upper extremity - Stroke Upper Limb Capacity Scale (SULCS) - administered by occupational therapist | Discharge (within 72 hours prior to discharge from inpatient rehabilitation unit - IRU)
  Measures upper limb capability in post-stroke patients. It includes basic upper limb capacity items (requiring little to no hand function) and advanced upper limb capacity items (necessitates moderate to good hand function). Includes 10 items related to daily activities of patient in the home environment; three items that test proximal upper limb (arm) capacity without the need for active wrist and finger movements; four items that test for upper limb capacity requiring basic control of wrist and finger movements; three items for upper limb capacity requiring advanced control of wrist and finger movements
Upper extremity - Upper Extremity Motricity Index - administered by occupational therapist | Discharge (within 72 hours prior to discharge from inpatient rehabilitation unit - IRU)
  Measures muscle strength of the paretic side of patient who has had a stroke. It includes three items: pinch grip, elbow flexion, shoulder abduction. Total scores range 0-100
Functional domain - Functional Independence Measure (FIM) - administered by various members of rehabilitation team (physical therapy, occupational therapy, nursing, speech therapist) | Discharge (within 72 hours prior to discharge from inpatient rehabilitation unit - IRU)
  A uniform system of measurement for disability. It measures the level of a patient's disability and indicates how much assistance is required for the individual to carry out activities of daily living.
Functional domain - Boston University Activity Measure for Post-Acute Care (AM-PAC) - administered by research assistant | Discharge (within 72 hours prior to discharge from inpatient rehabilitation unit - IRU)
  A questionnaire that examines a set of functional activities that are likely to be encountered by most adults during daily routines within the context of either an inpatient episode of care or outpatient post acute services. AM-PAC item banks are organized into three functional areas: Basic Mobility (101 items), Daily Activity (70 items), and Applied Cognitive (69 items).
Functional and cognitive domains - Executive Function Performance Test (EFPT) bill paying task - administered by occupational therapist | Discharge (within 72 hours prior to discharge from inpatient rehabilitation unit - IRU)
  An instrumental activities of daily living assessment (IADL) that tests the patient's ability to use five executive functions of a task: (1) initiation of a task, (2) organization, (3) sequencing, (4) safety and judgment, and (5) completion.

SECONDARY OUTCOMES:
Engagement in rehabilitation - Hopkins Rehabilitation Engagement Rating Scale (HRERS) - administered independently by occupational and physical therapists | Discharge (within 72 hours prior to discharge from inpatient rehabilitation unit - IRU)
  A 5-item clinician-rated measure to quantify the patient's engagement in acute rehabilitation services. The items are: frequency of the patient's rehabilitation attendance, frequency that the patient required verbal or physical prompts, frequency that the patient expressed positive attitude toward his rehabilitation activity, frequency that the patient acknowledged a need for rehabilitation, and frequency that the patient actively participated in the rehabilitation activity. Total score ranges 5-30, higher score represents greater engagement in therapy.
Cognition - Hopkins Verbal Learning Test-Revised (HVLT-R) - administered by speech therapist | Discharge (within 72 hours prior to discharge from inpatient rehabilitation unit - IRU)
  A brief verbal learning and memory test consisting of an exercise testing the patient's delayed recall.
Cognition - Trail Making Test (TMT) - administered by occupational therapist | Discharge (within 72 hours prior to discharge from inpatient rehabilitation unit - IRU)
  A 2-part test that provides information regarding attention, visual scanning, and executive function. Part A requires the participants to draw lines and connect 25 numbers scattered on a page. Part B requires that the participant connects the numbers and letters in order, alternating between letters and numbers
Cognition - Montreal Cognitive Assessment (MoCA) - administered by occupational therapist | Admission (within 72 hours after admission into the inpatient rehabilitation unit - IRU)
  A one-page instrument administered in 10 minutes for mild cognitive dysfunction in different cognitive domains. The MoCA Ranges from 0 to 30 points. The test assesses 8 domains of cognitive functioning: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.
Cognition - Digit Span test - administered by neuropsychologist | Discharge (within 72 hours prior to discharge from inpatient rehabilitation unit - IRU)
  A two-part assessment: Digits Forward and Digits Backward. Digits Forward primarily assesses short-term auditory memory while Digits Backward assesses the ability to manipulate verbal information in temporary storage. In Digits Forward, the subject listens to and repeats a sequence of numbers spoken aloud by the assessor. In Digits Backward, the subject listens to a sequence of numbers and repeats them in reverse order.
Cognition - Stroop Color and Word test - administered by neuropsychologist | Discharge (within 72 hours prior to discharge from inpatient rehabilitation unit - IRU)
  A five minute test of cognitive flexibility that assesses cognitive processing and provides diagnostic information on brain dysfunction and cognition. The Stroop Color and Word Test consists of a Word Page with color words printed in black ink, a Color Page with 'Xs' printed in color, and a color-Word Page with words from the first page printed in colors from the second page (the color and the word do not match). The subject reads words or names the ink colors as quickly as possible within a time limit.
Cognition - Logical memory test - administered by neuropsychologist | Discharge (within 72 hours prior to discharge from inpatient rehabilitation unit - IRU)
  Story A is read one time to the subject, who then orally provides any information recalled. Story B is read two times to the subject, with any recalled information provided after each reading. The neuropsychologist records the information recalled by the subject. After 30 minutes of other testing, the subject is asked to provide any information recalled from Story A and then Story B, and the assessor records this information. Fifteen yes/no recognition memory questions are then asked about each story and the recognition memory scores are recorded.
Cognition - Brief visuospatial memory test - administered by neuropsychologist | Discharge (within 72 hours prior to discharge from inpatient rehabilitation unit - IRU)
  A measure that consists of three Learning Trials. The subject views the stimulus page for 10 seconds (which displays six geometric figures) and is asked to draw as many of the figures as possible in the response booklet. A Delayed Recall Trial is administered after a 25-minute delay. A Recognition Trial, in which the subject is asked to identify which of 12 figures were included among the original geometric figures, is administered.
Cognition - Dementia Rating Scale - administered by neuropsychologist | Discharge (within 72 hours prior to discharge from inpatient rehabilitation unit - IRU)
  Assesses a patient's overall level of cognitive functioning. Consists of five subscales: Attention, Initiation/Perseveration, Construction, Conceptualization, and Memory. The most challenging tasks are presented first. If the first one or two tasks in a subscale are performed well, subsequent tasks in the subscale are marked as correct, and the assessor begins the next subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Michael O'Dell, MD, Principal Investigator — Weill Medical College of Cornell University; Joan Toglia, PhD, Study Director — Mercy College
Locations (1):
- New York Presbyterian/Weill Cornell Medical Center Rehabilitation Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mastrogiovanni, A., Toglia, J., & O'Dell, M. Relationship between Instrumental Activities of Daily Living (IADL) and Cognition after Mild Acute Stroke. Archives of Physical Medicine and Rehabilitation, 95(10), e12, 2014.
- [Background] Martinez, A. J., Fitzgerald, K. A., Mastrogiovanni, A. R., O'Dell, M. W., & Toglia, J. Exploring the Relationship of the Visuoexecutive Subscore of the Montreal Cognitive Assessment and Trails B to Functional Outcomes in Patients With Stroke. PM&R, 3(10): S162, 2011.
- [Background] Frantz, M.A.; Woznica, D., Schwabe, E.; Villanueva, M., Toglia, J., O'Dell, M. AM-PAC correlates with measures of impairment at discharge from inpatient stroke rehabilitation. American Journal of Physical Medicine & Rehabilitation: 93(3): a1-a97, 2014.
- [Background] O'Dell, M., Toglia, J., & Taub, M. Predicting Participation Level Six Month Following Inpatient Stroke Rehabilitation. Archives of Physical Medicine and Rehabilitation 10(96): e56, 2015.
- [Background] Tufaro, D. C., Toglia, J., O'Dell, M., & Villanueva, M. Concurrent Validity of the Stroke Upper Limb Capacity Scale (SULCS). Archives of Physical Medicine and Rehabilitation 10(95): e17, 2014.
- [Background] Parfene, C., Toglia, J., Taub, M., & O'Dell, M. W. Differences in identifying memory impairment using the Montreal Cognitive Assessment and Hopkins Verbal Learning Test-Revised delayed recall scores in an acute stroke population. Clinical Neuropsychologist 30(3): 393-394, 2016.
- [Background] Toglia J, Askin G, Gerber LM, Taub MC, Mastrogiovanni AR, O'Dell MW. Association Between 2 Measures of Cognitive Instrumental Activities of Daily Living and Their Relation to the Montreal Cognitive Assessment in Persons With Stroke. Arch Phys Med Rehabil. 2017 Nov;98(11):2280-2287. doi: 10.1016/j.apmr.2017.04.007. Epub 2017 May 4. PMID 28478128
- [Background] Taub, M., O'Dell, M., & Toglia, J. (2016). Relationship of Hopkins Rehabilitation Engagement Rating Scale to Baseline Cognition and FIM Change in Acute Inpatient Stroke Rehabilitation. Archives of Physical Medicine and Rehabilitation, 97(10), e111-e112.
- [Background] Meyer, A., Batistick, H., Toglia, J., Taub, M., & O'Dell, M. (2016). Factors Associated with a Large Time Differential Between Timed Up and Go and Gait Speed During Inpatient Stroke Rehabilitation. Archives of Physical Medicine and Rehabilitation, 97(10), e70-e71.
- [Derived] Lowder RJ, Jaywant A, Fridman CB, Toglia J, O'Dell MW. Cognitive impairment predicts engagement in inpatient stroke rehabilitation. Int J Rehabil Res. 2022 Dec 1;45(4):359-365. doi: 10.1097/MRR.0000000000000552. Epub 2022 Oct 17. PMID 36237146
- [Derived] O'Dell MW, Jaywant A, Frantz M, Patel R, Kwong E, Wen K, Taub M, Campo M, Toglia J. Changes in the Activity Measure for Post-Acute Care Domains in Persons With Stroke During the First Year After Discharge From Inpatient Rehabilitation. Arch Phys Med Rehabil. 2021 Apr;102(4):645-655. doi: 10.1016/j.apmr.2020.11.020. Epub 2021 Jan 10. PMID 33440132
- [Derived] Campo M, Toglia J, Batistick-Aufox H, O'Dell MW. Standardized Outcome Measures in Stroke Rehabilitation and Falls After Discharge: A Cohort Study. PM R. 2021 Mar;13(3):265-273. doi: 10.1002/pmrj.12396. Epub 2020 Jun 10. PMID 32358887
- [Derived] Jaywant A, Toglia J, Gunning FM, O'Dell MW. Subgroups Defined by the Montreal Cognitive Assessment Differ in Functional Gain During Acute Inpatient Stroke Rehabilitation. Arch Phys Med Rehabil. 2020 Feb;101(2):220-226. doi: 10.1016/j.apmr.2019.08.474. Epub 2019 Sep 10. PMID 31518565